CLINICAL TRIAL: NCT00246064
Title: The Infliximab Rheumatoid Arthritis Methotrexate Tapering (iRAMT) Protocol. Tapering Methotrexate in Patients With Rheumatoid Arthritis Beginning Therapy With Infliximab
Brief Title: The Infliximab Rheumatoid Arthritis Methotrexate Tapering (iRAMT) Protocol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centocor Ortho Biotech Services, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003127
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Infliximab infusions; Methotrexate; Remicade
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

INTERVENTIONS:
Drug: infliximab

SUMMARY:
The purpose of the study was to evaluate the ability of a maintenance dosage regimen of infliximab to achieve and sustain at least 40% improvement from baseline in the total joint count in patients with active Rheumatoid Arthritis (RA) during methotrexate tapering.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic autoimmune disorder of unknown etiology that occurs in approximately one percent of the population. Current therapy for RA comprises non-steroidal anti-inflammatory drugs (NSAIDs) in early stages of the disease, ultimately giving way to oral glucocorticoids and the disease-modifying anti-rheumatic drugs (DMARDs) as the disease progressively worsens. Therapy with DMARDs (e.g., D-penicillamine, auranofin, hydroxychloroquine, azathioprine, methotrexate) is not ideal in that they generally have a slow onset of action (measured in months), variable levels of effectiveness, and dose-limiting toxicity. Methotrexate (MTX) has become the DMARD of choice of many rheumatologists because of its faster mode of action and better record of prolonged use. However, despite the use of high doses of MTX, many patients only experience partial relief of symptoms and still have features of active disease. The current product labeling provides for a range of infliximab doses. Four fixed maintenance dose regimens proved to be safe and efficacious in the Anti-TNF Trial in Rheumatoid Arthritis with Concomitant Therapy (ATTRACT) trial. However, the efficacy of incremental dose titration in patients with RA who have not achieved or maintained a clinically important improvement from baseline status has not been established in a clinical trial setting. Additionally, whether MTX tapering is possible in those patients who have achieved a clinically important improvement from baseline status has not been demonstrated. The iRAMT trial utilizes a prescribed strategy for infliximab dose titration in the event that individuals do not achieve a 40% improvement in the combined swollen and tender joint count, or have a disease flare or recurrent worsening. The iRAMT trial defines a clinically important improvement as at least a 40% improvement from baseline. Once the 40% improvement is achieved, MTX tapering will be initiated as appropriate for the specific patient. The primary efficacy endpoint is the number (%) of patients on a maintenance dose of infliximab who achieve at least 40% improvement from baseline in the combined tender and swollen joint count and tolerate any reduction in MTX dose at Week 54. Hence, this trial will provide information regarding an infliximab dose titration strategy as well as a MTX tapering schedule in those patients responding to therapy. The iRAMT trial will examine, in a manner consistent with clinical practice, if a schedule of infliximab maintenance will allow for tapering of MTX to occur. Patients will receive Infliximab infusions at a minimum dose of 3 mg/kg at Weeks 0, 2, 6 and every 8 weeks thereafter until Week 46. During the study, the dose of infliximab may be increased by single 100-mg vials using a specified regimen up to a maximum of 10 mg/kg every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of RA according to the revised 1987 criteria of the American Rheumatism Association (Arnett et al., 1988)
* patients must have a minimum of 8 tender and 4 swollen joints with disease diagnosed at least 3 months prior to screening
* patients must have been using oral or parenteral MTX for at least the previous 3 months, and at a stable dose of 7.5 to 25 mg per week for at least the previous 1 month
* women of childbearing potential must test negative for pregnancy and be using adequate birth control measures
* patients must have a documented purified protein derivative (PPD) skin test performed at prescreening.

Exclusion Criteria:

* Patients who have received any prior treatment with infliximab or with any other therapeutic agent targeted at reducing tumor necrosis factor (TNF) (e.g., etanercept, pentoxifylline or thalidomide) within the previous 3 months
* patients who are incapacitated
* history of infected joint prosthesis within the previous 5 years
* patients with a concomitant diagnosis of congestive heart failure (CHF), history of or known malignancy within the previous 5 years, cases of active or latent tuberculosis (TB), acute or chronic serious infections within the past 3 months
* known substance abuse (drug or alcohol) within the previous 3 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2001-12; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the number (%) of patients on a maintenance dose of infliximab who achieve at least 40% improvement from baseline in the combined tender and swollen joint count and tolerate any reduction in MTX dose at Week 54

SECONDARY OUTCOMES:
Sustained improvement in signs and symptoms of RA at Week 54, as measured by the percentage improvement from baseline in ACR20 score. Improvement of the ACR20 core set components at Week 54.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Ortho Biotech Services, L.L.C. Clinical Trial, Study Director — Centocor Ortho Biotech Services, L.L.C.

REFERENCES:
- [Result] Fleischmann RM, Cohen SB, Moreland LW, Schiff M, Mease PJ, Smith DB, Keenan G, Kremer JM; iRAMT Study Group. Methotrexate dosage reduction in patients with rheumatoid arthritis beginning therapy with infliximab: the Infliximab Rheumatoid Arthritis Methotrexate Tapering (iRAMT) trial. Curr Med Res Opin. 2005 Aug;21(8):1181-90. doi: 10.1185/030079905X53261. PMID 16083527
- See also: The Infliximab Rheumatoid Arthritis Methotrexate Tapering (iRAMT) Protocol. Tapering Methotrexate in Patients with Rheumatoid Arthritis Beginning Therapy with Infliximab. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=128&filename=CR003127_CSR.pdf